CLINICAL TRIAL: NCT04585620
Title: Botulinum Toxin A as Treatment for Chronic Postsurgical Pain Following Lung Cancer Surgery: a Randomized Controlled Pilot Trial
Brief Title: Botulinum Toxin A as Treatment for Chronic Postsurgical Pain Following Lung Cancer Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allan Vestergaard Danielsen, MD (Other)
Responsible Party: Sponsor-Investigator, Allan Vestergaard Danielsen, MD, Principal Investigator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 74719
Record Dates: First submitted 2020-08-24; First posted 2020-10-14 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Pain; Post-thoracotomy Pain Syndrome; Pain, Neuropathic; Pain, Postoperative
Keywords: Botulinum toxin; Onabotulinum toxin A
MeSH Terms: conditions — Chronic Pain; Neuralgia; Pain, Postoperative | interventions — onabotulinum toxin A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BTX-A (Active Comparator): Onabotulinum toxin A is reconstructed with 4 ml of normal saline in a vial containing 100 U (Allergen Units).
  At a single treatment session, test subjects receive a series of subcutaneous injections with 2,5 U Onabotulinum toxin A equivalent to 0,1 ml of solution after reconstruction. One injection is given per 1 square centimeter in the painful area in relation to the scar on the chest wall. The maximum number of subcutaneous injections is 40, equivalent to a maximum dose of 100 U of Onabotulinum toxin in a total volume of 4 ml solution. The subcutaneous injections are administered using 26G 0.45 x 15 mm cannulae and 1 ml syringes.
  Interventions: Drug: Onabotulinum Toxin A
- Placebo (Placebo Comparator): At a single treatment session, test subjects receive a series of subcutaneous injections with one injection per 1 square centimeter in the painful area in relation to the scar on the chest wall with an inert solution, i.e. 0.1 ml injections of normal saline up to a total volume of 4 ml, depending on the area of the painful area. The subcutaneous injections are administered using 26G 0.45 x 15 mm cannulae and 1 ml syringes.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Onabotulinum Toxin A — Series of subcutaneous injections
  Other Names: BTX-A
  Arms: BTX-A
Drug: Normal saline — Series of subcutaneous injections
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Chronic postsurgical pain following lung cancer surgery is common with and 20-60 % develop chronic pain which persists more than six months after surgery. Causes and health impact of this pain have been comprehensively studied. Current treatment consists of combination of pain medication, physiotherapy and psychological therapy.

Botulinum Toxin A (BTX-A) has shown promising effects in a variety of chronic postsurgical pain syndromes. The use of BTX-A in lung cancer patients has only been presented in few case reports. No randomized controlled trials (RCT) have been executed to date.

Study objectives:

Determine recruitment potential among cured lung cancer patients with chronic postsurgical pain for an RCT and if the method of BTX-A administration is feasible and acceptable. Further more, this study will contribute to the stage testing of the hypothesis that chronic pain following thoracic surgery can be treated with BTX-A.

Methods:

Recruitment of test subjects:

Participiants are recruited among former lung cancer patients with chronic postsurgical pain, who have undergone radical treatment for lung cancer at the Department of Cardiothoracic Surgery, Aalborg University Hospital. Potential test subjects are invited by mail / e-mail.

Randomization and blinding:

Participants are randomized to receive a single series of subcutaneous injections with either Onabotulinum Toxin A (active agent) or inactive normal saline (Placebo) at the former operation site. Neither participant nor investigator will know which treatment is given until the end of the trial.

Data collection:

Data is collected by questionnaires delivered and answered by mail or digitally.

Data on the possible effects and possible adverse reactions are collected at multiple times until three months after treatment.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPP) following lung cancer surgery is common with an observed prevalence of 20-60 %. Causes and health impact have been comprehensively studied. Current treatment consists of combination of pain medication, physiotherapy and psychological therapy.

Botulinum Toxin A (BTX-A) has shown promising effects in a variety of chronic postsurgical pain syndromes. The use of BTX-A in lung cancer patients has only been presented in few case reports. No randomized clinical controlled trials (RCT) has been executed to date.

Study objectives:

Primary:

Determine recruitment potential among cured lung cancer patients with CPP for an RCT and if the method of BTX-A administration is feasible and acceptable to the test subjects.

Secondary:

Early stage testing of the hypothesis that CPP following thoracic surgery can be treated with this novel method.

Methods:

Recruitment of test subjects:

Test subjects are recruited among former lung cancer patients with chronic postsurgical pain, who have undergone radical treatment for lung cancer at the Department of Cardiothoracic Surgery, Aalborg University Hospital. Potential test subjects are invited by mail / e-mail.

Randomization and blinding:

Test subjects are randomized to receive a series of injections with either Onabotulinum Toxin A (active agent) or inactive normal saline (Placebo). Neither test subject nor investigator will know which treatment is given until the end of the trial.

Experimental treatment:

The investigator examines the skin area of the test subject at the operation site and performs a sensory examination with pin prick and sensory brush. The area is located and marked and divided into quadrants of one square centimeter. An area of maximum 40 square centimeters is marked.

At a single treatment session, test subjects receives either active agent or placebo through a series of subcutaneous injections. One injection is given in each marked quadrant of the treatment area. The maximal number of injections is 40.

Follow-up:

After the treatment, test subjects report pain symptoms and intensity, use of pain medication and occurrence of adverse events weekly.

After 30 and 90 days after treatment more comprehensive and additional data is collected concerning neuropathic symptoms, activities of daily life, general health and level of function.

Data collection Data is collected by questionnaires delivered to test subjects by mail or digitally.

Endpoints:

Primary:

1. Recruitment of 30 test subjects.
2. Half of the first half of included test subject must complete the treatment.
3. Half of test subjects in total mus complete the treatment.

Secondary:

1. Pain at rest, coughing and when active Numerical rating score (NRS) for presence of pain before and after treatment and course of pain symptoms.
2. General Health Short form 36 Health Survey on physical, social and mental level of function on a score from 0 to 100.
3. Neuropathic Pain Symptoms Inventory (NPSI) NRS
4. Activities of daily life Impact and intensity of pain categorically in 16 situations of daily life.
5. Patient's Global Impression of Change (PGIC) Rating of global change perceived by the test subject from "More Worse" to "Much better" and a scale from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 18 years of age or above.
2. Patients who have undergone pulmonary surgery because of suspicion or confirmed pulmonary malignancies.
3. Patients who are radically treated for pulmonary malignancy
4. Patients who suffers from chronic pain or unpleasant sensation at the site of scar at least six months after surgery with fully healed surgical wounds.

Exclusion Criteria:

1. Patients who cannot understand oral and written information.
2. Patients who were not radically operated.
3. Patients with other concomitant or other active cancer diseases.
4. Patients with chronic pain in the chest wall prior to surgery.
5. Pregnant women or women planning to get pregnant in the study period.
6. Patients with autoimmune neuromuscular diseases, sclerosis, peripheral neuromuscular disturbances and general muscle weakness or atrophy.
7. Patients with intolerance or allergy to BOTOX®.
8. Patients who are at present treated with BTX-A or similar neuromuscular blocking drug or have received such in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 12 months
  Recruitment of 30 test subjects within twelve months.
Incidence of treatment procedure disruption | 12 months
  Proportion of test subjects terminating the treatment procedure after randomization by request due to unacceptable pain or discomfort during the procedure.

SECONDARY OUTCOMES:
Neuropathic Pain Symptoms Inventory (NPSI) | Baseline, 1 and 3 moths after treatment
  Numeric Rating Scale, range 0 (no pain) to 10 (worst pain imaginable) in whole numbers
Activities of daily life | Baseline, 1 and 3 months
  Impact and intensity of pain categorically in 16 situations of daily life. Categorically reported as "Avoid", "Major restriction", "Some restriction", "Minor restriction", "No restriction" or "Do not perform"
Patient's Global Impression of Change (PGIC) | 1 and 3 months after treatment.
  Rating of global change perceived by the test subject from "More Worse" to "Much better" and a scale from 0 to 10.
Pain at rest, coughing and when active | Weekly after treatment for three months
  Numeric Rating Scale, range 0 (no pain) to 10 (worst pain imaginable) in whole numbers
General Health | Baseline, 1 and 3 months after treatment
  Short form 36 Health Survey on physical, social and mental level of function on a score from 0 to 100.
Pain at procedure | Baseline
  Evaluation of pain/discomfort at administration of BTX-A using subcutaneous injection in the skin of the chest wall. Numeric Rating Scale, range 0 (no pain) to 10 (worst pain imaginable) in whole numbers

OTHER OUTCOMES:
Incidence of treatment procedure disruption for the first half of test subjects | Through study inclusion period of 12 months
  Half of the first half of included test subject must complete the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Allan V Danielsen, MD, Principal Investigator — Dept. of Cardiothoracic Surgery, Aalborg University Hospital
Locations (1):
- Dept. of Cardiothoracic Surgery, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No